CLINICAL TRIAL: NCT03655496
Title: Patient-centred Home-based Management of Heart Failure
Acronym: PACEMAN-HF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CareLigo AB (Industry)
Collaborators: Karolinska University Hospital (Other); Danderyd's hospital (Unknown); Stockholm South General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PACEMAN-HF
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
Keywords: patient centred; m-health; e-health; home-based; self-care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Subject to standard care.
- Intervention group (Experimental): Exposed to the home-based tool.
  Interventions: Device: Home-based tool

INTERVENTIONS:
Device: Home-based tool — The tool consists of a tablet computer and a Bluetooth connected weight scale. The patient is encouraged to use the tool daily. The weight is titrates the dose of diuretics and a short tip about how to improve living with heart failure, this is presented on the screen. Every five days the patient assess their self-perceived symptoms on the tablet computer. If the weight increases by 2kg or more in 3 days or less, the high dose is recommended for two days, after which the effect on the weight is assessed. If the weight increased was reverted, the dose is returned to normal and if it is still elevated, an alert on the table computer. If the self-assessed symptoms deteriorate, the same type of alert will appear on screen, urging the patient to contact the health care provider.
  Arms: Intervention group

SUMMARY:
A novel home-based tool for self-management is to be evaluated for heart failure patients. The tool assists the patient with symptom monitoring, education and titration of diuretics. Patients who were recently hospitalized for heart failure will be randomized to receiving the tool or standard care for six months. The primary end-point will be self-care behaviour, as measured with the validated instrument the European Heart failure self-care behaviour Scale 9-item questionnaire (Jaarsma et al). Secondary end-points are in-hospital days due to heart failure, quality of life (general and disease-specific) as measured by the SF-36 and KCCQ questionnaires, and finally knowledge about heart failure, assessed by the Dutch Heart Failure Knowledge Scale.

DETAILED DESCRIPTION:
Patients who are admitted to the emergency unit for decompensated heart failure at the three largest clinics in Stockholm, Sweden, are screened for recruitment. For patients to be eligible for study participation, they shall be discharged from the hospital to the general practitioner without being referred to a nurse led heart failure clinic, which is considered the gold standard in terms of improving patients' self-care behaviour. At the point of discharge, patients are approached about study participation and those who accept will be provided study information and forced to provide a written consent to participate. Continuous sampling is employed. Baseline characteristics are noted, as well as baseline data collected for the following end-points: Self-care, using the European Heart Failure Self-care Behaviour Scale (EHFScB), general quality of life using the SF-36 questionnaire, disease-specific quality of life using the Kansas City Cardiomyopathy Questionnaire (KCCQ) and knowledge about heart failure using the Dutch Heart Failure Knowledge Scale (DHFKS). After this data is collected patients will be randomized, using sealed envelopes, to either receive standard care or receive the home-based tool that constitutes the intervention investigated. Within one week after discharge, the patients randomized to the intervention group will have he tool installed in their home.

The tool consists of a tablet computer locked to a specialized software, and a Bluetooth connected weight scale. Every day the patient is encouraged by the tablet computer to step up on the weight scale. The weight is wirelessly transferred to the tablet computer and today's dose of diuretics is shown on screen together with a short tip about how to improve living with heart failure. Every five days the patient assess their self-perceived symptoms, as prompted on the tablet computer. For every patient equipped with the tool, a patient-specific normal dose of diuretics, as well as a high dose is input in the tool at the point of randomization. If the weight increases by 2kg or more in 3 days or less, the high dose is recommended for two days, after which the effect on the weight is assessed. If the weight was decreased back to where it was prior to the rapid weight gain, the dose is returned to normal and if it is still elevated, the patient will be encouraged to call his/her health care provider at the number presented on the table computer. If the self-assessed symptoms deteriorate, the same type of warning will appear on screen, urging the patient to contact the health care provider. Both the intervention patients and the control patients will be given the same discharge information in writing, describing the most important parts of self-management for heart failure patients. The data collected at baseline will be collected again after 3 months and 6 months after randomization. After 6 months data about hospitalizations will be retrieved from the medical records and adjudicated as either heart failure-hospitalization or not. The adjudication will be done by the cardiologists participating in the study and as the focus of the study is in estimating the net/marginal incidence rate ratio of in-patient hospitalization, absorbing competing events (e.g. death) will be handled by censoring.

ELIGIBILITY:
Inclusion Criteria:

* admitted due to acute heart failure
* diagnosed heart failure according to European Society of Cardiology (ESC) guidelines 2012
* prescribed loop-diuretics
* Signed letter of consent

Exclusion Criteria:

* more than mild cognitive impairment
* pregnancy
* having attended nurse-led heart failure clinic the past 12 months, or referred to one following this current hospitalization
* life-expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2013-12-18 (Actual); Study Completion 2013-12-18 (Actual)

PRIMARY OUTCOMES:
Self-care behaviour | 6 months
  Assessed by the validated instrument European Heart Failure Self-care Behaviour Scale. It measures how well the patient adheres to advice provided from the health care professional. It si made up of nine questions to which the patient answers between "completely agree" and "completely disagree", corresponding to a score of 1 or 5 respectively. The possible scores on the questionnaire range from 9 to 45, where 9 corresponds to the most desireable self-care behaviour and 45 to the least favourable.

SECONDARY OUTCOMES:
In-hospital days due to heart failure | 6 months
  Data retrieved from the medical records after the intervention period is completed. All hospitalizations analyzed and adjudicated as either heart failure related or not.
Quality of life (general) | 6 months
  Assessed by the 36-item Short Form survey (SF-36). The instrument includes 8 multi-item scales plus a single-item scale to compare the patient's current health with that 1 year ago. The 8 domains are physical functioning, physical role, bodily pain, general health vitality, social functioning, role of emotional health and role of mental health. SF-36 also consists of two summary scores: mental and physical. The scores range from 0 to 100 and higher scores indicate better quality of life.
Quality of life (disease-specific) | 6 months
  Assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ). KCCQ is a 23-item (15 questions), self-administrating,disease-specifi c instrument that quantifi es 6 domains (scales) and 2 summary scores of patients' health status. The 6 domains are physical limitations, symptom score, symptom change, self-effi cacy, social interference and QoL. The 2 summary scores are labelled: clinical summary scores and overall summary scores. All scale scores are transformed to 0 - 100 scale, in which a higher score indicates better health related quality of life (HRQoL).
Knowledge about heart failure | 6 months
  Assessed by the Dutch Heart Failure Knowledge Scale (DHFKS), which consists of 15 multiple-choice items (0 - 15). It measures knowledge in HF in general, symptom recognition and treatment. Higher scores indicate more knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Hagerman, PhD, Principal Investigator — Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hagglund E, Lynga P, Frie F, Ullman B, Persson H, Melin M, Hagerman I. Patient-centred home-based management of heart failure. Findings from a randomised clinical trial evaluating a tablet computer for self-care, quality of life and effects on knowledge. Scand Cardiovasc J. 2015 Aug;49(4):193-9. doi: 10.3109/14017431.2015.1035319. Epub 2015 Jun 4. PMID 25968968
- [Background] Melin M, Hagglund E, Ullman B, Persson H, Hagerman I. Effects of a Tablet Computer on Self-care, Quality of Life, and Knowledge: A Randomized Clinical Trial. J Cardiovasc Nurs. 2018 Jul/Aug;33(4):336-343. doi: 10.1097/JCN.0000000000000462. PMID 29369123
- [Derived] Hovland-Tanneryd A, Melin M, Hagglund E, Hagerman I, Persson HE. From randomised controlled trial to real world implementation of a novel home-based heart failure tool: pooled and comparative analyses of two clinical controlled trials. Open Heart. 2019 May 28;6(1):e000954. doi: 10.1136/openhrt-2018-000954. eCollection 2019. PMID 31217992